CLINICAL TRIAL: NCT07361237
Title: A Phase l Clinical Study to Evalute the Safety,Tolerability,Pharmacokinetic Characteristics,and Preliminary Anti-tumor Efficacy of HJ-004-02 Tablets in Patients With Non-squamous Non-small Cell Lung Cancer With Epidermal Growth Factor Receptor (EGFR) Mutations
Acronym: HJ-004-02-101
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Caicun Zhou, chief physician, Tongji University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTR20254077
Record Dates: First submitted 2025-12-17; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HJ-004-02-101 (Experimental)
  Interventions: Drug: HJ-004-02 tablets

INTERVENTIONS:
Drug: HJ-004-02 tablets — Single dose: Fasting, oral administration, as a single dose, taken with warm water. Multiple doses: Fasting, oral administration, as a single dose, taken with warm water, once daily (dosing frequency may be adjusted based on study data), with 28 days as one cycle.

SUMMARY:
Single dose: Fasting, oral administration, as a single dose, taken with warm water. Multiple doses: Fasting, oral administration, as a single dose, taken with warm water, once daily (dosing frequency may be adjusted based on study data), with 28 days as one cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged >=18 years and <75 years
2. Clinical diagnosis of NSCLC.
3. Subjects must have experienced disease progression after standard therapy, or be intolerant to or unsuitable for standard therapy, or have no available standard therapy.
4. Subjects must provide 3-5 archived tumor tissue slides
5. Subjects must have non-squamous NSCLC with one or more positive EGFR mutations
6. At least one measurable lesion according to RECIST v1.1 (In Phase Ia, lesions that are assessable but not measurable are acceptable).
7. ECOG performance status score of 0-1
8. Life expectancy >=12 weeks.
9. (1) Hematologic Function:Absolute neutrophil count (ANC) >= 1.5×10^9/L;Platelet count (PLT) >= 100×10^9/L;Hemoglobin (HGB) >=9.0 g/dL; (2)Hepatic Function:Total bilirubin (TBIL) <=1.5 × upper limit of normal (ULN) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) For those without liver metastases, <=2.5 × ULN, orFor those with liver metastases, <=5 × ULN; (3)Renal Function:Creatinine <=1.5 × ULN; if >1.5 × ULN, creatinine clearance ≥50 mL/min [Creatinine clearance calculated using the Cockcroft-Gault formula (see Appendix 2: Cockcroft-Gault Formula)] (4)Coagulation Panel Note: For subjects receiving anticoagulant therapy, the investigator will determine whether the international normalized ratio (INR) and activated partial thromboplastin time (APTT) are within a safe therapeutic range. INR <= 1.5×ULN;APTT <= 1.5×ULN.
10. Contraception is required during the trial period.

Exclusion Criteria:

1. Within the four weeks prior to the administration of HJ-004-02 tablets, the patient had received other anti-tumor treatments such as biological therapy, immunotherapy, radiotherapy, and chemotherapy.
2. Participation in an investigational drug study with treatment or use of an investigational device within 4 weeks before the first dose of HJ-004-02 tablets. 3. Anticipated need for any other form of anti-tumor therapy during the study.

4. Toxicity from prior therapy has not resolved to <=Grade 1 according to NCI-CTCAE v5.0 criteria, with the exception of alopecia and long-term stable chronic disease.

5. Presence of histological transformation, and ALK, HER2, KRAS, ROS1, FGFR, NTRK, RET, BRAF gene abnormalities in EGFR-TKI non-dependent drug resistance; 6. History of severe eye disorder prior. 7. History of severe dermatosis prior. 8. Subjects who have gastrointestinal disease 9. Subjects who have received treatment with P-gp inhibitors, potent CYP3A4 inhibitors 10. Subjects with uncontrolled pleural effusion, ascites, or pericardial effusion requiring repeated drainage procedures, as judged by the investigator.

11. Subjects with symptomatic brain metastasis, metastases to meninges, or spinal cord compression.

12. Subjects with an active infection of >=Grade 2 13. Subjects with a history of allergy to the active ingredient or inactive excipients of HJ-004-02 tablets, or to drugs with a similar chemical structure or class to HJ-004-02 tablets.

14. Subjects with a confirmed immunodeficiency disease, and/or a positive HIV test result at screening.

15. Subjects with active hepatitis B 16. Subjects with positive syphilis antibodies and a positive titer test. 17. Active tuberculosis. 18. Presence of a malignancy other than the indication of this study within <=5 years before the first dose of HJ-004-02 tablets 19. Subjects who have had a clinically significant cerebrovascular disorder within 6 months before the first dose of HJ-004-02 tablets, 20. Subjects who have undergone major surgery or severe traumatic injury within 4 weeks before the first dose of HJ-004-02 tablets, or who are expected to require major surgery during the study.

21. History of interstitial lung disease (ILD) 22. Subjects with any haemorrhagic diathesis or coagulopathy 23. Subjects with a known psychiatric illness 24. Those who have received a live attenuated vaccine within 28 days before the first dose of the investigational product or plan to receive one during the study and within 60 days after the end of investigational product treatment.

25. Female subjects who are pregnant or breastfeeding. 26. Any other condition that, in the investigator's judgment, would hinder the subject's participation in the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
AE | through study completion, an average of 1 year
  Incidence and severity of adverse events (AEs)
DLT | at the end of cycle1（each cycle is 28 days）
  Incidence of dose-limiting toxicities (DLTs) during the DLT observation period

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No